CLINICAL TRIAL: NCT00554099
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of a 12 Week Treatment of Acute Diverticulitis With Asacol® 2.4 g/Day (400 mg Mesalamine Tablet), Followed by a 9 Month Treatment-free Observation Period
Brief Title: Asacol Acute Diverticulitis(DIVA)Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007020
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Mesalamine; Probiotics; Nutrition Assessment; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Days 1 thru Days 10 to 14 (Visit 2): daily antibiotic therapy, dietary advice, and 6 placebo tablets (matching mesalamine) once a day. Visit 2 thru Week 12 : 1 placebo capsule (matching probiotic) and 6 placebo tablets (matching mesalamine) daily.
  Interventions: Drug: Placebo; Other: Dietary Advice; Drug: Antibiotic for Diverticulitis
- Mesalamine (Active Comparator): Days 1 thru 10-14 (Visit 2): daily antibiotic therapy, dietary advice and 6 - 400 mg mesalamine tablets once a day. Visit 2 thru Week 12: 1 placebo capsule (matching probiotic) and 6 - 400 mg mesalamine tablets daily.
  Interventions: Drug: Mesalamine; Other: Dietary Advice; Drug: Antibiotic for Diverticulitis
- Mesalamine & Probiotic (Active Comparator): Days 1 thru 10-14 (Visit 2): daily antibiotic therapy, dietary advice and 6 - 400 mg mesalamine tablets once daily. Visit 2 thru Week 12: 1- Bifidobacterium infantis 35624 capsule and 6 - 400 mg mesalamine tablets daily
  Interventions: Drug: Probiotic; Other: Dietary Advice; Drug: Antibiotic for Diverticulitis

INTERVENTIONS:
Drug: Mesalamine — 6 - 400 mg tablets once daily
  Arms: Mesalamine
Drug: Probiotic — Once capsule daily Bifidobacterium infantis 35624 added at Visit 2 (Day 10 + 4 days)
  Other Names: Align
  Arms: Mesalamine & Probiotic
Drug: Placebo — 6 placebo tablets for first 10 (+4) days followed by once daily placebo tablets.
  Arms: Placebo
Other: Dietary Advice — Dietary advice
Drug: Antibiotic for Diverticulitis — Physician recommended antibiotic for Diverticulitis taken for 10-14 days. Antibiotic not specified for study.

SUMMARY:
The purpose of this study is to determine whether Asacol® 2.4 g/day (400 mg Mesalamine) is safe and effective in the treatment of diverticulitis.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of Asacol® 2.4 g/day in generally healthy, adult patients who have had an attack of acute diverticulitis. The study will evaluate the safety and efficacy of a 12 week treatment with Asacol® followed a 9 month non-treatment observation period in approximately 180 patients with acute diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of acute diverticulitis
* Female patients must be postmenopausal (at least 1 year without spontaneous menses) or surgically sterile or have a negative urine pregnancy test and practice acceptable contraception (e.g., abstinence; oral, intramuscular, or implanted hormonal contraception [at least 3 months prior to enrollment]; 2-barrier methods [e.g., condom, diaphragm, or spermicide]; intrauterine device or verbal report of partner with history of non-reversed vasectomy)
* Willing and able to participate in the study and provide a signed informed consent

Exclusion Criteria:

* Presence of diverticular complications (e.g., fistula, abscess, obstruction, stenosis);
* Active or recent history (within 6 months) of a peptic ulcer;
* Prior history of irritable bowel syndrome (IBS), as determined by the Investigator;
* History of major abdominal surgery (as determined by the Investigator);
* History of GI surgery within 3 months of diagnosis of acute diverticulitis;
* History of immunocompromising disease, human immunodeficiency virus (HIV) infection, or acquired immunodeficiency syndrome (AIDS);
* If female patient, active or recent history of endometriosis or dysmenorrhea;
* Received a dose of a product that contains, or is metabolized to, mesalamine by any route within 4 weeks before the screening visit;

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Balske, MD, PhD, Study Director — Procter and Gamble
Locations (36):
- United States (36):
  - Research Site, Tucson, Arizona
  - Research Facility, Los Angeles, California
  - Research Site, Merced, California
  - Research Site, Oakland, California
  - Research Facility, Orange, California
  - Research Site, Palm Springs, California
  - Research Site, Pasadena, California
  - Research Site, Lafayette, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Jacksonsville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Winter Park, Florida
  - Research Facility, Zephyrhills, Florida
  - Research Site, Pratt, Kansas
  - Research Site, Monroe, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Chesterfield, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Mexico, Missouri
  - Research Facility, Cedar Knolls, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Lake Success, New York
  - Research Site, Setauket, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Facility, Harrisburg, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cranston, Rhode Island
  - Research Site, Longview, Texas
  - Research Site, Odessa, Texas
  - Research Site, Chesapeake, Virginia
  - Research Facility, Monroe, Wisconsin

REFERENCES:
- [Derived] Stollman N, Magowan S, Shanahan F, Quigley EM; DIVA Investigator Group. A randomized controlled study of mesalamine after acute diverticulitis: results of the DIVA trial. J Clin Gastroenterol. 2013 Aug;47(7):621-9. doi: 10.1097/MCG.0b013e31828003f6. PMID 23426454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient screened 6 Dec 2007
Pre-assignment Details: Randomization 1:1:1 ratio with subsequent stratification based on number of prior episodes (1 attack vs. more than 1 attack).
Groups:
- Placebo: Placebo tablets (matching mesalamine, 6 tablets daily)
- Mesalamine: 400 mg mesalamine (6 tablets daily)
- Mesalamine & Probiotic: 400 mg mesalamine (6 tablets daily) plus Align (1 capsule daily)
Period: Treatment Period (12 Weeks)
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Started | 41 | 40 | 36
Completed | 29 | 32 | 27
Not Completed | 12 | 8 | 9
Not completed — Adverse Event | 3 | 5 | 1
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Recurrent diverticulitis,surgery require | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 4
Period: Non-Treatment Phase (9 Months)
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Started | 29 | 32 | 27
Completed | 22 | 27 | 24
Not Completed | 7 | 5 | 3
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Relapse | 2 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic | Total
Number analyzed (Participants) | 41 | 40 | 36 | 117
Age, Customized [Number; unit: Participants]
  < 65 years | 31 | 28 | 25 | 84
  >= 65 years | 10 | 12 | 11 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 19 | 61
  Male | 22 | 17 | 17 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 4 | 10
  Not Hispanic or Latino | 37 | 38 | 32 | 107
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 39 | 39 | 33 | 111
  Black | 2 | 0 | 2 | 4
  Asian (Oriental) | 0 | 0 | 1 | 1
  Multi-racial | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 36 | 117

OUTCOME MEASURES:

1. Primary Outcome: Global Symptom Score (GSS) at Week 12, Primary Efficacy Population
Description: GSS - Abdominal Pain & Symptom Rating, scale 0-none (better) to 6-severe (worse) for each of the following categories: abdominal pain, abdominal tenderness, nausea/vomiting, bloating, constipation, diarrhea, mucus in stool, feeling urge to evacuate but no bowel movement, painful straining with bowel movement, pain/difficulty urinating. Total minimum score 0 (better), total maximum score 60 (worse).
Time Frame: 12 Weeks
Population: Primary Efficacy Population - Subset of ITT population including only patients with GSS value at Week 12 and baseline GSS of at least 12.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 41 | 40 | 36
Scores on a Scale | 7.3 (1.30) | 4.4 (1.07) | 5.9 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; It was assumed that the placebo treatment group and mesalamine treatment group would have an average composite score of 8.4 and 5.88 at Week 12, respectively. The common standard deviation was set to 4.5 based on the 2 standard deviation rule. Based on these assumptions, 60 patients per treatment group required to detect 30% treatment difference at 1-sided, 0.1 level of significance, with 80% power; Test type: Superiority or Other; p = 0.3781, ANCOVA; Fixed effects for treatment, number of diverticulitis attacks and baseline value as covariate; Mean Difference vs. Placebo = -3.0, 90% CI 1-sided [upper limit -0.809], Standard Error of Mean 1.69
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6285, ANCOVA; Fixed effects for treatment, number of diverticulitis attacks and baseline value as covariate; Mean Difference vs. Placebo = -1.4, 90% CI 1-sided [upper limit 0.815], Standard Error of Mean 1.74
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4365, ANCOVA; Fixed effects for treatment, number of diverticulitis attacks and baseline value as covariate; Mean Difference vs. Asacol = 1.6, 90% CI 1-sided [upper limit 3.573], Standard Error of Mean 1.58

2. Secondary Outcome: Percentage of Responders at Week 12 - ITT Population
Description: Responder - patient whose GSS scores for all symptoms were either 0 or 1 GSS - Abdominal Pain & Symptom Rating, scale 0-none (better) to 6-severe (worse) for each of the following categories: abdominal pain, abdominal tenderness, nausea/vomiting, bloating, constipation, diarrhea, mucus in stool, feeling urge to evacuate but no bowel movement, painful straining with bowel movement, pain/difficulty urinating. Total minimum score 0 (better), total maximum score 60 (worse).
Time Frame: 12 Weeks
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 41 | 40 | 36
Percentage of Participants | 41.4 | 62.5 | 48.1
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; Test type: Superiority or Other; p = 0.0576, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = 21.1, 90% CI 1-sided [lower limit 5.1], Standard Error of Mean 12.53
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.3248, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = 6.8, 90% CI 1-sided [lower limit -10.2], Standard Error of Mean 13.27
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.8596, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Mesalamine = -14.4, 90% CI 1-sided [lower limit -30.8], Standard Error of Mean 12.87

3. Secondary Outcome: Percentage of Responders at Week 52 - ITT Population
Description: as for outcome 2
Time Frame: 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 29 | 32 | 27
Percentage of Participants | 50.0 | 66.7 | 29.2
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; Test type: Superiority or Other; p = 0.1266, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = 16.7, 90% CI 1-sided [lower limit -1.3], Standard Error of Mean 14.00
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.9288, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = -20.8, 90% CI 1-sided [lower limit -38.9], Standard Error of Mean 14.13
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.9962, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = -37.5, 90% CI 1-sided [lower limit -54.1], Standard Error of Mean 12.98

4. Secondary Outcome: Change in GSS From Baseline to Week 12 - ITT Population
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 41 | 40 | 36
Scores on a Scale | -16.14 (2.082) | -17.63 (1.825) | -16.11 (2.110)
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; Test type: Superiority or Other; p = 0.3082, ANOVA; Fixed effects for treatment and number of diverticulitis attacks; LS Mean Difference vs. Placebo = -1.400, 90% CI 1-sided [upper limit 2.196], Standard Error of Mean 2.784
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.5113, ANOVA; Fixed effects for treatment and number of diverticulitis attacks; LS Mean Difference vs. Placebo = 0.083, 90% CI 1-sided [upper limit 3.832], Standard Error of Mean 2.903
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.6988, ANOVA; Fixed effects for treatment and number of diverticulitis attacks; LS Mean Difference vs. Mesalamine = 1.483, 90% CI 1-sided [upper limit 5.145], Standard Error of Mean 2.836

5. Secondary Outcome: Change in GSS From Baseline to Week 52 - ITT Population
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: ITT Population
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 29 | 32 | 27
Scores on a Scale | -16.82 (2.527) | -17.30 (2.040) | -16.00 (1.931)
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; Test type: Superiority or Other; p = 0.4448, ANOVA; Fixed effects for treatment and number of diverticulitis attacks; LS Mean Difference vs. Placebo = -0.428, 90% CI 1-sided [upper limit 3.541], Standard Error of Mean 3.067
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.6029, ANOVA; Fixed effects for treatment and number of diverticulitis attacks; LS Mean Difference vs. Placebo = 0.825, 90% CI 1-sided [upper limit 4.903], Standard Error of Mean 3.151
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.6615, ANOVA; Fixed effects for treatment and number of diverticulitis attacks; LS Mean Difference vs. Mesalamine = 1.253, 90% CI 1-sided [upper limit 5.129], Standard Error of Mean 2.996

6. Secondary Outcome: Withdrawal Due to Surgery for Diverticulitis, Percentage, ITT Population, Week 12
Time Frame: 12 Weeks
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 41 | 40 | 36
Percentage of Participants | 2.4 | 5.0 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; Test type: Superiority or Other; p = 0.7165, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = 2.6, 90% CI 1-sided [upper limit 7.9], Standard Error of Mean 4.20
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.1708, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = -2.4, 90% CI 1-sided [upper limit 0.6], Standard Error of Mean 2.41
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.1039, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Mesalamine = -5.0, 90% CI 1-sided [upper limit -0.6], Standard Error of Mean 3.45

7. Secondary Outcome: Recurrent Diverticulitis, Percentage, ITT Population, Week 12
Description: At least one report of recurrent diverticulitis since the last visit (prior to the Week 12 visit).
Time Frame: 12 Weeks
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 41 | 40 | 36
Percentage of Participants | 20.0 | 12.5 | 11.8
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; Test type: Superiority or Other; p = 0.1907, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = -7.5, 90% CI 1-sided [upper limit 3.0], Standard Error of Mean 8.21
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.1730, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = -8.2, 90% CI 1-sided [upper limit 2.5], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.4613, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Mesalamine = -0.7, 90% CI 1-sided [upper limit 9.0], Standard Error of Mean 7.61

8. Secondary Outcome: Recurrent Diverticulitis, Percentage, ITT Population, Week 52
Description: At least one report of recurrent diverticulitis since the last visit (prior to the Week 52 visit).
Time Frame: 52 Weeks
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Number analyzed (Participants) | 29 | 32 | 27
Percentage of Participants | 31.0 | 28.1 | 37.0
Statistical Analysis 1: Comparison: Placebo vs Mesalamine; Test type: Superiority or Other; p = 0.3983, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = -2.9, 90% CI 1-sided [upper limit 12.1], Standard Error of Mean 11.70
Statistical Analysis 2: Comparison: Placebo vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.6721, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Placebo = 6.0, 90% CI 1-sided [upper limit 22.2], Standard Error of Mean 12.66
Statistical Analysis 3: Comparison: Mesalamine vs Mesalamine & Probiotic; Test type: Superiority or Other; p = 0.7703, Cochran-Mantel-Haenszel; Stratified by number of diverticulitis attacks; Difference vs. Mesalamine = 8.9, 90% CI 1-sided [upper limit 24.6], Standard Error of Mean 12.23

ADVERSE EVENTS:
Time Frame: 6 Dec 2007 thru 1 Mar 2010
Description: Intent to Treat Population. Adverse Events were differentiated by occurring either in the treatment period (initial 12 weeks therapy) or the non-treatment period (9 month follow up period) using the corresponding numbers from participant flow for each of the trial periods specified.
Arm/Group | Placebo | Mesalamine | Mesalamine & Probiotic
Serious Adverse Events (participants affected / at risk) | 6/41 | 5/40 | 0/36
Other Adverse Events (participants affected / at risk) | 32/41 | 37/40 | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=41) | Mesalamine (N=40) | Mesalamine & Probiotic (N=36)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial Thrombosis Limb (Vascular disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Atrioventricular Block (Cardiac disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Bronchopneumonia (Infections and infestations) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon Operation (Surgical and medical procedures) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0/29 (0) | 1/32 (1) | 0/27 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=41) | Mesalamine (N=40) | Mesalamine & Probiotic (N=36)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 12 (14) | 4 (5)
Abdominal Pain Lower (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1/29 (1) | 1/32 (1) | 0/27 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anal Pruritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/29 (1) | 1/32 (1) | 0/27 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (3)
Bartholin's Cyst (Reproductive system and breast disorders) | 0/29 (0) | 0/32 (0) | 1/27 (1)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Blood Urea Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1/29 (1) | 1/32 (1) | 0/27 (0)
C-Reactive Protein Increased (Investigations) | 1/29 (1) | 1/32 (1) | 1/27 (1)
Clostridial Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 0/29 (0) | 0/32 (0) | 1/27 (1)
Colonic Polyp (Gastrointestinal disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (4) | 3 (3)
Coronary Artery Disease (Cardiac disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (7) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulum Intestinal (Gastrointestinal disorders) | 0/29 (0) | 0/32 (0) | 1/27 (1)
Dyslipidaemia (Investigations) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Dyspepsia (Gastrointestinal disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Feeling Abnormal (General disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0/29 (0) | 0/32 (0) | 1/27 (1)
Fungal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Gastroenteritis Viral (Infections and infestations) | 1/29 (1) | 1/32 (1) | 1/27 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1/29 (1) | 1/32 (1) | 0/27 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Investigations) | 1/29 (1) | 0/32 (0) | 1/27 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1/29 (1) | 0/32 (0) | 1/27 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Joint Sprain (Injury, poisoning and procedural complications) | 0/29 (0) | 0/32 (0) | 1/27 (1)
Liver Function Test Abnormal (Investigations) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Localized Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1/29 (2) | 0/32 (0) | 0/27 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0/29 (0) | 0/32 (0) | 1/27 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Oedema (General disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Perirectal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3/29 (3) | 1/32 (1) | 2/27 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rash Generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Sciatica (Nervous system disorders) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0/29 (0) | 0/32 (0) | 1/27 (1)
Sinusitis (Infections and infestations) | 0/29 (0) | 1/32 (1) | 1/27 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue Dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1/29 (1) | 1/32 (1) | 2/27 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1/29 (1) | 0/32 (0) | 0/27 (0)
Vaginal Infection (Infections and infestations) | 0/29 (0) | 1/32 (1) | 0/27 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less